CLINICAL TRIAL: NCT00479024
Title: CARE (Visipaque 320 and Isovue 370 in Cardiac Angiography in REnally Impaired Patients); FOLLOW-UP STUDY
Brief Title: Follow-up Study to Previous CARE Trial
Status: Completed | Type: Observational
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Steven Sireci, Executive Director, Corporate medical Support, Bracco Diagnostics, Inc.
Other Study IDs: IOP112
Record Dates: First submitted 2007-05-23; First posted 2007-05-25 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Moderate to Severe Chronic Kidney Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observation: patients enrolled in previous trial IOP 104; collecting clinical outcome data on these same patients
  Interventions: Drug: iodinated contrast agent

INTERVENTIONS:
Drug: iodinated contrast agent — iodinated contrast agent either 370 stength of iopamidol or 320 strength of visipaque

SUMMARY:
To determine comparative 1-year outcomes in renally impaired patients who previously underwent cardiac angiography with Isovue®-370 or Visipaque™ 320 as part of the IOP-104 trial protocol and were evaluable for determination of post-contrast significant renal injury (defined as >25% increase in SCr or >25% increase in cystatin C).

ELIGIBILITY:
Inclusion Criteria: (from previous CARE trial)

* • Screening eGFR between 20 and 59 mL/min/1.73m2

  * Baseline SCr obtained within 72 hours and before hydration or, if obtained after hydration started, had the screening blood sample obtained within 72 hours of contrast administration
  * At least one post dose blood sample available
  * Received randomized contrast agent
  * Underwent only one cardiac angiography procedure (diagnostic cardiac angiography followed by PCI was considered as one procedure if confirmed by investigator and total duration does not exceed 12 hours), then for this study
  * Provides written Informed Consent and is willing to comply with protocol requirements;
  * Was included in the patient list provided by Bracco;
  * At least 1 year has passed since the patient's participation ended in the original CARE trial, as determined from the list provided by Bracco

Exclusion Criteria:

* • Screening eGFR outside the range of 20 and 59 mL/min/1.73m2

  * Unstable kidney disease or requiring dialysis upon enrollment
  * Prior to the post-dose blood draw, suffered a critical clinical event that would affect the reliability of serological measurement of renal function
  * Did not receive randomized contrast agent per CARE protocol
  * Did not undergo a cardiac angiography procedure per CARE protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Sireci, M.D., Study Chair — Bracco Diagnostics, Inc
Locations (1):
- Cardiovascular Associates, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Solomon RJ, Mehran R, Natarajan MK, Doucet S, Katholi RE, Staniloae CS, Sharma SK, Labinaz M, Gelormini JL, Barrett BJ. Contrast-induced nephropathy and long-term adverse events: cause and effect? Clin J Am Soc Nephrol. 2009 Jul;4(7):1162-9. doi: 10.2215/CJN.00550109. Epub 2009 Jun 25. PMID 19556381